CLINICAL TRIAL: NCT07280221
Title: WEgovy Real World Assessment of Weight Loss in Korea (WE-WALK): a Multi-centre, Prospective, Single-arm, Nonintervention Study to Investigate the Effectiveness and Safety of Once-weekly Semaglutide 2.4 mg for People Living With Obesity in Routine Clinical Practice in Korea
Brief Title: WEgovy Real World Assessment of Weight Loss in Korea
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9536-7850; U1111-1306-1595 (Other: WHO)
Record Dates: First submitted 2025-11-24; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Once weekly Wegovy: Participants will be treated with commercially available semaglutide. The treating physician will initiate treatment with commercially available semaglutide prior to and independently from the decision to include the participant in the study.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Semaglutide injection will be self-administered once weekly subcutaneously.

SUMMARY:
This study is to investigate the effectiveness and safety of Wegovy (semaglutide) in Korean patients living with obesity in routine clinical practice. The purpose of this study is to investigate the change in body weight and other clinical characteristics related to body weight in patients living with obesity. Participants will be treated with Wegovy (semaglutide) as prescribed by their doctor, in accordance with normal clinical practice. The study will last for about 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. The decision to initiate treatment with commercially available Wegovy (semaglutide) has been made by the patient and the treating physician before and independently from the decision to include the patient in this study.
3. Initiating treatment with Wegovy (semaglutide) for the first time and according to locally approved label.
4. Male or female, aged ≥ 19 years at the time of signing the informed consent.

Exclusion Criteria:

1. Previous participation in clinical studies including treatment with Wegovy (semaglutide). Participation is defined as providing informed consent in a previous study.
2. Female patient who is pregnant, breast-feeding, or intends to become pregnant and is of childbearing potential not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice).
3. Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be treated with commercially available semaglutide. The treating physician will initiate treatment with commercially available semaglutide prior to and independently from the decision to include the participant in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight | From baseline (week 0) to 24 weeks
  Percent (%)

SECONDARY OUTCOMES:
Absolute change in body weight | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Kilogram (kg)
Percentage change in body weight | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Percent (%)
Achievement in body weight reduction more than or equal to (≥) 5% | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Count of patients
Achievement in body weight reduction ≥ 10% | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Count of patients
Achievement in body weight reduction ≥ 15% | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Count of patients
Achievement in body weight reduction ≥ 20% | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Count of patients
Change in body composition of Lean body mass | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Kg
Change in body composition of Total fat mass | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Kg
Change in body composition of Lean body mass | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Percent (%)
Change in body composition of Total fat mass | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Percent (%)
Change in Body mass index (BMI) | From baseline (week 0) up to 8, 16, 24, 32, 40, 52 weeks
  Kilogram per meter square (kg/m^2)
Change in the proportion of patients by BMI Class I obesity (25 to 29.9 kg/m^2) | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Count of patients
Change in the proportion of patients by BMI Class II obesity (30 to 34.9 kg/m^2) | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Count of patients
Change in the proportion of patients by BMI Class III obesity (≥35 kg/m^2) | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Count of patients
Change in waist circumference | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Centimetre (cm)
Change in cardiometabolic parameters - Systolic blood pressure (SBP) | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Millimetres of mercury (mmHg)
Change in cardiometabolic parameters - Diastolic blood pressure (DBP) | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  mmHg
Change in cardiometabolic parameters - Fasting plasma glucose (FPG) | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Milligram per deciliter (mg/dL)
Change in cardiometabolic parameters - Haemoglobin A1c (HbA1c) | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  Percent (%)
Change in cardiometabolic parameters - Lipids: total cholesterol (TCh) | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  mg/dL
Change in cardiometabolic parameters - Lipids: high-density lipoprotein cholesterol (HDL-C) | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  mg/dL
Change in cardiometabolic parameters - Lipids: low-density lipoprotein cholesterol (LDL-C) | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  mg/dL
Change in cardiometabolic parameters - Lipids: triglycerides (TG) | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  mg/dL
Change in cardiometabolic parameters - Lipids: free fatty acid (FFA) | From baseline (week 0) to 8, 16, 24, 32, 40, 52 weeks
  mg/dL
Change in status of type two diabetes mellitus (T2DM) | Baseline (week 0) to 52 weeks [or end of the study (EOS)]
  Count of patients
Change in status of Hypertension | Baseline (week 0) to 52 weeks (or EOS)
  Count of patients
Change in status of Dyslipidemia | Baseline (week 0) to 52 weeks (or EOS)
  Count of patients
Number of treatment-emergent adverse events (TEAEs) | From baseline (week 0) to 52 weeks (or EOS)
  Count of events
Number of serious TEAEs | From baseline (week 0) to 52 weeks (or EOS)
  Count of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Daejeon Endo Internal Medicine Clinic, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com